CLINICAL TRIAL: NCT00002402
Title: Phase I/II Trial to Evaluate the Safety and Immunogenicity of AIDSVAX B/B and B/E Vaccines in the United States
Brief Title: A Study of AIDSVAX B/B and AIDSVAX B/E, Two Possible Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VaxGen (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Prevention
Other Study IDs: VAX 002
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-08

CONDITIONS: HIV Infections
Keywords: HIV-1; Dose-Response Relationship, Drug; Acquired Immunodeficiency Syndrome; AIDS Vaccines; HIV Seronegativity; Antigens, Viral; Alum Compounds
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Aluminum Hydroxide

INTERVENTIONS:
Biological: MN rgp120/HIV-1 and GNE8 rgp120/HIV-1
Biological: MN rgp120/HIV-1 and A244 rgp120/HIV-1
Biological: Aluminum hydroxide

SUMMARY:
The purpose of this study is to see if it is safe and effective to give AIDSVAX B/B or AIDSVAX B/E, two potential HIV vaccines, to HIV-negative volunteers.

DETAILED DESCRIPTION:
Patients are randomized to 1 of the 2 following arms and administered 1 or 2 injections into the deltoid muscle at 0, 1, 6, and 12 months:

Arm A: Patients receive 1 of 3 doses of AIDSVAX B/B vaccine (MN rgp120/HIV-1 plus GNE8 rgp120/HIV-1) in alum adjuvant.

Arm B: Patients receive AIDSVAX B/E (MN rgp120/HIV-1 plus A244 rgp120/HIV-1) vaccine in alum adjuvant.

Patients are evaluated at 1 hr, 3 days, and 14 days after each immunization and at 18 months after the first immunization.

An interim analysis is performed after all patients receive the second dose (at 1 month).

ELIGIBILITY:
Patients must:

Be HIV-uninfected men and women at low or intermediate risk for HIV-1 infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Dr Frank Judson / Director of Public Health Dept, Denver, Colorado
  - Johns Hopkins Bloomberg School of Public Health, Washington D.C., District of Columbia
  - Fenway Community Health Ctr, Boston, Massachusetts
  - Saint Louis Univ Health Sciences Ctr, St Louis, Missouri

REFERENCES:
- [Background] Mayer K, Judson F, Gorse G, Harro C, Peterson M, Zaharias E, Good J, Shibata R, Lee S, Eastman D, Chernow M, Francis D, Berman P. A phase I/II trial to evaluate the safety and immunogenicity of the AIDSVAX B/B vaccine in the United States (final report). 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 178)